CLINICAL TRIAL: NCT07401719
Title: EFFECTS OF MODIFIED CLAMSHELL EXERCISES ON PAIN, RANGE OF MOTION AND FUNCTIONAL OUTCOMES IN PATIENTS WITH HIP OSTEOARTHRITIS GRADE Ⅱ
Brief Title: Effects of Modified Clamshell Exercises in Patients With Hip Osteoarthritis Grade II.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCPT/DPT/ERB/44
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteo Arthritis of Hip
Keywords: Modified Clamshell Exercises; Hip Osteoarthritis Grade II; Hip Osteoarthritis; Clamshell Exercises; Hip Disability and Osteoarthritis Outcome Score (HOOS-12) scale; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: This study follows a randomized controlled trial (RCT) design to compare the effectiveness of modified clamshell exercises and clamshell exercises, each combined with conventional hip osteoarthritis exercises, in patients with Grade II hip osteoarthritis. Eligible participants will be randomly allocated into three parallel groups using a computer-generated randomization sequence to ensure balanced group assignment. The first group will receive modified clamshell exercises in combination with conventional exercises, the second group will receive clamshell exercises with conventional exercises, and the third group will receive conventional exercises only. A double-blinded approach will be used, in which both the participants and outcome assessors will be blinded to group allocation. Outcomes will be assessed at baseline and at 3, 6, and 12 weeks to evaluate changes in pain intensity, hip function, and range of motion. This study design allows for a controlled comparison of exercise-based
Who Masked: Participant, Outcomes Assessor
Masking Description: This study uses a double-blinded design. Participants and outcome assessors will be blinded to group allocation to minimize performance and selection bias. Group assignment will be concealed using sealed, opaque, sequentially numbered envelopes. All outcome assessments, including pain intensity, hip function, and range of motion, will be performed by an independent outcome assessor who will remain blinded to group allocation throughout the study. Due to the nature of exercise-based interventions, the treating therapists will not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Modified Clamshell Exercise (Experimental): This group will receive modified clamshell exercises along with conventional exercises.
  Interventions: Other: Modified clamshell exercise; Other: Conventional exercises
- Clamshell exercise (Experimental): Participants in this group will receive clamshell exercises along with conventional exercises.
  Interventions: Other: Clamshell Exercises; Other: Conventional exercises
- Conventional Exercises (Active Comparator): This group will only receive conventional exercises including TENS, hot pack, bridging, sideways hip lifts, standing hip extension, and double hip rotation exercises.
  Interventions: Other: Conventional exercises

INTERVENTIONS:
Other: Modified clamshell exercise — This group will receive modified clamshell exercises along with conventional exercises. Time for each session will be 40 minutes. Patient will receive 3 sessions a weeks for 12 weeks.
  Arms: Modified Clamshell Exercise
Other: Clamshell Exercises — This group will receive Clamshell exercises along with conventional exercises. Each session will last for 40 minutes. Patient will receive 3 sessions a weeks for 12 weeks.
  Arms: Clamshell exercise
Other: Conventional exercises — This group will only receive conventional exercises including TENS, hot pack bridging, sideways hip lifts, standing hip extension and double hip rotation. time of each session will be 40 minutes. Patient will receive 3 sessions a weeks for 12 weeks.

SUMMARY:
This study focuses on patients diagnosed with Grade II hip osteoarthritis, a degenerative joint condition characterized by pain, reduced range of motion, muscle weakness, and functional limitations. Hip osteoarthritis is commonly assessed using the Kellgren-Lawrence (KL) classification system, with Grade II representing definite osteophyte formation with possible joint space narrowing, where conservative management is strongly recommended. Exercise therapy, particularly strengthening of the hip abductor muscles, plays a key role in improving pelvic stability, reducing pain, and enhancing functional outcomes. Clamshell exercises are widely used to activate the gluteus medius and minimus muscles, while modified clamshell exercises are designed to optimize muscle recruitment and reduce compensatory movements.

A total of 54 participants with Grade II hip osteoarthritis will be included in the study and allocated into three groups. Group A will receive clamshell exercises along with conventional exercise therapy, Group B will receive modified clamshell exercises in addition to conventional exercise therapy, and Group C will receive a conventional exercise program alone. Pain intensity will be assessed using the Visual Analog Scale (VAS), which ranges from 0 to 10. Hip joint range of motion will be measured using a goniometer, and functional outcomes will be evaluated using the Hip Disability and Osteoarthritis Outcome Score-12 (HOOS-12). The aim of this study is to compare the effects of clamshell exercises, modified clamshell exercises, and conventional exercise programs to determine the most effective intervention for reducing pain, improving hip joint range of motion, and enhancing functional outcomes in patients with Grade II hip osteoarthritis.

DETAILED DESCRIPTION:
Hip osteoarthritis (OA) is a chronic degenerative joint disorder characterized by progressive deterioration of articular cartilage, changes in subchondral bone, osteophyte formation, and narrowing of the joint space. These structural changes lead to pain, stiffness, reduced range of motion, muscle weakness, gait abnormalities, and functional limitations, ultimately affecting mobility, independence, and quality of life. Hip osteoarthritis is a common musculoskeletal condition, particularly in middle-aged and older adults, with global prevalence estimates indicating that approximately 5-10% of adults over the age of 45 are affected. Mechanical factors such as altered joint biomechanics, abnormal load distribution across the hip joint, femoroacetabular impingement, repetitive joint loading, previous trauma, and weakness of surrounding musculature play a significant role in the development and progression of the disease.

Radiographic assessment is commonly used to classify the severity of hip osteoarthritis, with the Kellgren-Lawrence (KL) grading system being the most widely accepted. The KL classification ranges from Grade 0 to Grade IV. Grade 0 indicates no radiographic evidence of osteoarthritis. Grade I shows doubtful joint space narrowing with possible osteophyte formation. Grade II is characterized by definite osteophyte formation with possible joint space narrowing. Grade III includes multiple moderate osteophytes, definite joint space narrowing, sclerosis, and possible bony deformity. Grade IV represents severe osteoarthritis with large osteophytes, marked joint space narrowing, severe sclerosis, and definite bony deformity. Grade II hip osteoarthritis represents an early stage of the disease in which conservative management is strongly recommended to reduce symptoms, improve function, and slow disease progression.

Exercise therapy is a core component of conservative management for hip osteoarthritis and plays a vital role in improving muscle strength, joint stability, range of motion, and overall functional performance. Strengthening of the hip abductor muscles is particularly important, as these muscles contribute to pelvic stability and optimal load transfer during functional activities such as walking and stair climbing. Clamshell exercises are commonly prescribed to activate and strengthen the gluteus medius and minimus muscles. Modified clamshell exercises involve changes in positioning or execution to enhance muscle recruitment, improve neuromuscular control, and minimize compensatory movements, potentially resulting in improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

- (1) Patients between 45 to 60 years. (2) Both male and female patients with hip osteoarthritis grade II were selected for this study.

(3) Patients with Hip Osteoarthritis grade II. (4) Patients with pain more than 6 months.

Exclusion Criteria:

* (1) Patients with Cardiac disorders. (2) Patient with other current lower extremity pathologies (e.g., peripheral vascular disease, septic arthritis) (3) Patients with low back surgery.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 12 weeks
  Pain intensity will be assessed using the Visual Analog Scale (VAS). The VAS is a widely used, valid, and reliable subjective measure of pain intensity, where participants rate pain on a scale from 0 to 10 . A score of 0 means no pain, while 10 represent worst imaginable pain. Participants. The VAS is sensitive to changes over time and is commonly used in clinical and research settings to evaluate treatment effectiveness. Pain intensity will be assessed at baseline, 3 weeks, 6 weeks, and 12 weeks
ROM | 12 weeks
  Range of motion (ROM) of the hip joint will be assessed using a universal goniometer. Goniometric measurement is a standard and objective clinical method used to evaluate joint mobility and functional movement in individuals with hip osteoarthritis. Hip abduction, and external rotation will be measured following standardized positioning and measurement procedures to ensure consistency and reliability. Goniometric ROM measurements provide quantitative data to identify movement limitations, monitor functional improvements, and assess the effectiveness of therapeutic exercise interventions. ROM assessments will be performed at baseline, 3 weeks, 6 weeks, and 12 weeks.

SECONDARY OUTCOMES:
Functional Outcomes | 12 weeks
  Functional outcome will be assessed using the Hip Disability and Osteoarthritis Outcome Score-12 (HOOS-12). The HOOS-12 is a validated, patient-reported outcome measure designed to evaluate hip-related symptoms, pain, and functional limitations in individuals with hip osteoarthritis. It consists of 12 items covering key domains of hip function and quality of life. Each item is scored on a Likert scale, and scores are transformed to a 0-100 scale, with higher scores indicating better hip function and fewer symptoms. The HOOS-12 is sensitive to clinical changes and suitable for both short-term and long-term assessment of functional improvement. Functional outcomes will be measured at baseline, 3 weeks, 6 weeks, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Principal investigator, Principal Investigator — Ghurki Trust and Teaching Hospital
Locations (1):
- Ghurki Trust and Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Exercise Therapy Program in Rehabilitation of Patients with Primary Hip Osteoarthritis
- [Background] Exercise in patients with hip osteoarthritis-effects on muscle and functional performance
- [Background] Kaleem S, Noor R, Bashir MS, Ikram M. Effects of clamshell exercises in terminal extension lag after ACL reconstruction.
- [Background] Effect of modified clamshell exercise on gluteus medius, quadratus lumborum and anterior hip flexor in participants with gluteus medius weakness